CLINICAL TRIAL: NCT03552393
Title: An Open-Label, Single-Arm, Multicenter Study to Ascertain the Optimal Starting Dose of MIRCERA® Given Subcutaneously for the Maintenance Treatment of Anemia in Pediatric Patients With Chronic Kidney Disease on Dialysis or Not Yet on Dialysis.
Brief Title: Ascertain the Optimal Starting Dose of Mircera Given Subcutaneously for Maintenance Treatment of Anemia in Pediatric Patients With Chronic Kidney Disease on Dialysis or Not Yet on Dialysis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NH19708; 2016-004779-39 (EudraCT Number)
Record Dates: First submitted 2018-04-27; First posted 2018-06-11 (Actual); Results first posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Anemia; Renal Insufficiency, Chronic
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mircera (Experimental): Mircera will be administered subcutaneously once every 4 weeks
  Interventions: Drug: Mircera

INTERVENTIONS:
Drug: Mircera — The initial dose of Mircera will be one of nine starting doses corresponding to the prefilled syringe strengths based on the total weekly erythropoiesis-stimulating agent (ESA) dose during the screening period.
  Other Names: Methoxy polyethylene glycol-epoetin beta

SUMMARY:
Ascertain the starting dose of Mircera given subcutaneously for the maintenance treatment of anemia in pediatric participants with chronic kidney disease (CKD) on dialysis or not yet on dialysis when switching from stable subcutaneous (SC) maintenance treatment with epoetin alfa, epoetin beta, or darbepoetin alfa.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric participants 3 months to 17 years of age with clinically stable chronic renal anemia
* CKD with estimated glomerular filtration rate (eGFR) of < 45 mL/min/1.73 m2 (determined by the Bedside Schwartz formula) or dialysis treatment for at least 8 weeks before the first dose of Mircera
* For participants on peritoneal dialysis (PD): a weekly Kt/V≥ 1.8
* For participants on hemodialysis (HD): adequate HD, urea reduction ratio (URR) > 65% or Kt/V > 1.2 for participants on HD three times per week.

Participants with fewer than or more than three HD sessions per week should have a weekly Kt/V≥ 3.6.

* Baseline Hb concentration 10.0-12.0 g/dL determined from the mean of two Hb values measured at Visit 1 (Week -3) and Visit 2 (Week -1)
* Stable SC maintenance treatment with epoetin alfa, epoetin beta, or darbepoetin alfa with the same dosing interval for at least 6 weeks before the first dose of Mircera
* Stable dose of epoetin alfa, epoetin beta, or darbepoetin alfa treatment with no weekly dose change > 25% (increase or decrease) for at least 4 weeks before the first dose of Mircera
* Adequate iron status defined as ferritin≥100 ng/mL or transferrin saturation (TSAT)≥ 20% (or percentage of hypochromic red cells < 10%); mean of two values measured during screening.

Exclusion Criteria:

* Overt gastrointestinal bleeding within 8 weeks before screening or during the screening period
* RBC transfusions within 8 weeks before screening or during the screening period
* Hemoglobinopathies (e.g., homozygous sickle-cell disease, thalassemia of all types) Hemolytic anemia, Active malignant disease
* PD subjects with an episode of peritonitis within the past 30 days prior to screening and/or during the screening period
* Uncontrolled or symptomatic inflammatory disease (e.g., systemic lupus erythematosus)
* Uncontrolled hypertension as assessed by the investigator
* Epileptic seizures within 3 months prior to screening and during the screening period
* Administration of any investigational drug within 4 weeks prior to screening or planned during the study
* Severe hyperparathyroidism (intact parathyroid hormone [PTH]≥ 1000 pg/mL or whole PTH≥ 500 pg/mL) or biopsy-proven bone marrow fibrosis
* Kidney transplant with use of immunosuppressive therapies known to exacerbate anemia
* Known hypersensitivity to recombinant human erythropoietin (EPO), polyethylene glycol, or any constituent of the study drug formulation
* Anti-EPO antibody (AEAB)-mediated pure red cell aplasia (PRCA) or history of AEAB mediated PRCA or positive AEAB test result in the absence of PRCA
* High likelihood of early withdrawal or interruption of the study (e.g., planned living donor kidney transplant within 5 months of study start)
* Planned elective surgery during the entire study period

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- United States (7):
  - University of Alabama at Birmingham; Pediatric Nephrology, Birmingham, Alabama
  - Loma Linda University health, Loma Linda, California
  - Emory University School of Med; Pediatrics, Atlanta, Georgia
  - Children'S Mercy Hospital; Pediatric Nephrology, Kansas City, Missouri
  - RWJBarnabas Health, West Orange, New Jersey
  - East Carolina University; Brody School of Medicine, Greenville, North Carolina
  - UT Southwestern Medical Center; Pediatrics Dept., Dallas, Texas
- France (3):
  - Hopital Jeanne De Flandre; Pediatrie, Lille
  - Gh Necker Enfants Malades; Nephrologie, Paris
  - Höpital Hautepierre; Pediatrie 1, Strasbourg
- Hungary (2):
  - Semmelweis University; 1st Department of Pediatrics, Pediatric Nephrology Center, Budapest
  - Debreceni Egyetem Klinikai Központ; Gyermekklinika, Debrecen
- Italy (2):
  - Clinica Pediatrica II De Marchi, Milan, Lombardy
  - Ospedale Infantile Regina Margherita; U.O. Autonoma di Nefrologia, Dialisi e Trapianto, Turin, Piedmont
- Vilnius University Children's Hospital, Vilnius, Lithuania
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne; Klinika Chorob Nerek i Nadciśnienia Dzieci i Mlodziezy, Gdansk
  - Uniwersytecki Szpital Dziecięcy w Krakowie; Oddz.Nefrologii i Nadciśnienia Tętniczego/Stacja Dializ, Krakow
  - Instytut "Centrum Zdrowia Matki Polki; Klinika Pediatrii i Immunologii i Nefrologii, Lodz
  - Szpital Specjalistyczny dla Dzieci i Doroslych; Oddzial Kliniczny Pediatrii i Nefrologii, Torun
  - Szpital Kliniczny nr 1 im. prof. Szyszko; Oddz. Nefrologii Dzieciecej z Pododdziałem Dializoterapii, Zabrze
- Spain (2):
  - Hospital Universitari Vall d'Hebron; Servicio de Nefrologia, Barcelona
  - Hospital Universitario Virgen del Rocio; Servicio de Nefrologia Pediatrica, Seville

REFERENCES:
- [Derived] Warady BA, Meyer Reigner S, Tirodkar C, Drozdz D. Subcutaneous C.E.R.A. for the Maintenance Treatment of Anemia in Pediatric Patients With CKD: A Phase 2, Open-Label, Single-Arm, Multicenter Study. Am J Kidney Dis. 2023 Jun;81(6):684-694.e1. doi: 10.1053/j.ajkd.2022.11.006. Epub 2022 Dec 29. PMID 36587890

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The core study was 23 weeks and consisted of three periods: screening (3 weeks), dose titration (16 weeks) and evaluation (4 weeks). Participants completing the 20 weeks of treatment with hemoglobin (Hb) within +/- 1g/dL of their baseline and within the target range of 10-12 g/dL were eligible to enter an optional 24-week safety extension period.
Pre-assignment Details: A total of 40 pediatric participants (ages 3 months to 17 years) with a diagnosis of anemia due to chronic kidney disease (CKD) who may or may not have been on dialysis at the time of study start were switched from stable subcutaneous (SC) maintenance treatment with epoetin alfa/beta or darbepoetin to methoxy polyethylene glycol-epoetin beta (Mircera).
Groups:
- Mircera: Mircera was administered subcutaneously once every 4 weeks.
Period: Core Period
Arm/Group | Mircera
Started | 40
Completed | 38
Not Completed | 2
Not completed — Kidney Transplant | 1
Not completed — Prohibited Medication | 1
Period: Safety Extension Period
Arm/Group | Mircera
Started | 25
Completed | 21
Not Completed | 4
Not completed — Kidney Transplant | 4

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population included all participants enrolled in the study.
Arm/Group | Mircera
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.32 (5.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 30
  More than one race | 0
  Unknown or Not Reported | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin (Hb) Concentration Between the Baseline and the Evaluation Period for Each Patient
Description: The Hb change from baseline was calculated on a per-participant basis using an individual's average for both the baseline and evaluation periods and taking the difference. The baseline period was defined as the time between the day of first study dose and the previous 35 days. The evaluation period was defined as the period between Week 17 and Week 21, inclusive.
Time Frame: Baseline up to Week 21
Population: ITT population included all participants enrolled in the study. Number analyzed is the number of participants with Hb concentration assessment at specified time points.
Measure: Mean (Standard Deviation); unit: grams/deciliter (g/dL)
Arm/Group | Mircera
Number analyzed (Participants) | 38
grams/deciliter (g/dL)
  Baseline | 11.05 (0.51)
  Change at Evaluation Period | 0.48 (1.03)

2. Secondary Outcome: Number of Participants With an Average Hb Concentration During the Evaluation Period Within ± 1 g/dL of Their Baseline Hb and Above, Within or Below the Range of 10-12 g/dL
Description: Number of participants with an average Hb concentration during the evaluation period within ± 1 g/dL of their baseline Hb is reported as well as the number of participants with an average Hb concentration above, within or below the range of 10-12 g/dL. The evaluation period was defined as the period between Week 17 and Week 21 inclusive.
Time Frame: Week 17 up to Week 21
Population: ITT population included all participants enrolled in the study. Hb values within 21 days after blood transfusion(s) were excluded from analysis. Number analyzed is the number of participants with Hb concentration assessment at specified time points.
Measure: Number; unit: participants
Arm/Group | Mircera
Number analyzed (Participants) | 38
participants
  Hb Above 1 g/dL of Baseline | 15
  Hb Maintained Within ± 1 g/dL of Baseline | 19
  Hb Below 1 g/dL of Baseline | 4
  Hb Above 12 g/dL | 12
  Hb Maintained Within 10-12 g/dL | 24
  Hb Below 10 g/dL | 2

3. Secondary Outcome: Mean Hb Values and Change From Baseline
Description: The mean Hb concentration over time and the mean change in Hb from baseline over time are presented.
Time Frame: Baseline, Weeks 3, 5, 9, 13, 17, 19, 21, 25, 29, 33, 37, 41, 45
Population: ITT population included all participants enrolled in the study. Number analyzed signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Mircera
Number analyzed (Participants) | 40
g/dL
  Baseline | 11.02 (0.53)
  Week 3 | 11.69 (0.97)
  Change at Week 3 | 0.67 (0.74)
  Week 5 | 11.21 (1.02)
  Change at Week 5 | 0.19 (0.94)
  Week 9: number analyzed (Participants) | 39
  Week 9 | 11.68 (1.42)
  Change at Week 9: number analyzed (Participants) | 39
  Change at Week 9 | 0.64 (1.21)
  Week 13: number analyzed (Participants) | 38
  Week 13 | 11.56 (1.17)
  Change at Week 13: number analyzed (Participants) | 38
  Change at Week 13 | 0.51 (1.10)
  Week 17: number analyzed (Participants) | 37
  Week 17 | 11.46 (1.33)
  Change at Week 17: number analyzed (Participants) | 37
  Change at Week 17 | 0.42 (1.39)
  Week 19: number analyzed (Participants) | 37
  Week 19 | 11.81 (1.11)
  Change at Week 19: number analyzed (Participants) | 37
  Change at Week 19 | 0.77 (1.14)
  Week 21: number analyzed (Participants) | 38
  Week 21 | 11.10 (0.91)
  Change at Week 21: number analyzed (Participants) | 38
  Change at Week 21 | 0.05 (0.99)
  Week 25: number analyzed (Participants) | 25
  Week 25 | 11.29 (1.04)
  Change at Week 25: number analyzed (Participants) | 25
  Change at Week 25 | 0.21 (1.12)
  Week 29: number analyzed (Participants) | 23
  Week 29 | 11.22 (1.18)
  Change at Week 29: number analyzed (Participants) | 23
  Change at Week 29 | 0.15 (1.11)
  Week 33: number analyzed (Participants) | 24
  Week 33 | 11.09 (1.11)
  Change at Week 33: number analyzed (Participants) | 24
  Change at Week 33 | 0.02 (1.24)
  Week 37: number analyzed (Participants) | 24
  Week 37 | 11.04 (0.77)
  Change at Week 37: number analyzed (Participants) | 24
  Change at Week 37 | -0.03 (0.90)
  Week 41: number analyzed (Participants) | 22
  Week 41 | 10.83 (0.83)
  Change at Week 41: number analyzed (Participants) | 22
  Change at Week 41 | -0.22 (1.03)
  Week 45: number analyzed (Participants) | 21
  Week 45 | 10.68 (1.02)
  Change at Week 45: number analyzed (Participants) | 21
  Change at Week 45 | -0.35 (1.13)

4. Secondary Outcome: Change in Mircera Dose Over Time
Description: A dose change was defined as a change in the administered dose strength compared to the preceding dose.
Time Frame: Week 1 to Week 17
Population: Safety population included all participants who received at least one dose of study drug regardless of whether they withdrew prematurely or not. Number analyzed signifies number of participants evaluable at specified time points.
Measure: Median (Full Range); unit: micrograms (µg)
Arm/Group | Mircera
Number analyzed (Participants) | 40
micrograms (µg)
  Week 1 | 75.00 [15.0 to 360.0]
  Week 5: number analyzed (Participants) | 39
  Week 5 | 75.00 [15.0 to 360.0]
  Change at Week 5: number analyzed (Participants) | 39
  Change at Week 5 | 0.00 [-50.0 to 75.0]
  Week 9: number analyzed (Participants) | 39
  Week 9 | 50.00 [0.0 to 360.0]
  Change at Week 9: number analyzed (Participants) | 39
  Change at Week 9 | 0.00 [-250.0 to 190.0]
  Week 13: number analyzed (Participants) | 38
  Week 13 | 50.00 [0.0 to 360.0]
  Change at Week 13: number analyzed (Participants) | 38
  Change at Week 13 | -25.00 [-120.0 to 210.0]
  Week 17: number analyzed (Participants) | 38
  Week 17 | 50.00 [0.0 to 250.0]
  Change at Week 17: number analyzed (Participants) | 38
  Change at Week 17 | -20.00 [-250.0 to 120.0]

5. Secondary Outcome: Ratio of Mircera Starting Dose (Week 1) to the Dose at Week 17
Description: The ratio of Mircera dose was calculated as the median (min-max) ratio of starting dose (Week 1) to the dose at Week 17. Participants who withdrew before Week 17 or who were not administered a Mircera dose at Week 17 visit due to the applicable dose adjustment rules were excluded from the ratio computation.
Time Frame: Week 1, Week 17
Population: Participants who received a dose of study drug on Week 1 and Week 17 were included in the analysis.
Measure: Median (Full Range); unit: ratio
Arm/Group | Mircera
Number analyzed (Participants) | 33
ratio | 1.44 [0.2 to 3.8]

6. Secondary Outcome: Number of Participants With Adverse Events by Severity as Assessed by Highest World Health Organization (WHO) Toxicity Grade
Description: An adverse event is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product, any new disease, or exacerbation of existing disease (a worsening in the character, frequency, or severity of a known condition), recurrence of an intermittent medical condition or any deterioration in a laboratory value or other clinical test.
Time Frame: Baseline up to Week 45
Population: Safety population included all participants who received at least one dose of study drug regardless of whether they withdrew prematurely or not.
Measure: Number; unit: participants
Arm/Group | Mircera
Number analyzed (Participants) | 40
participants
  Grade 1-2 | 25
  Grade 3-4 | 8

7. Secondary Outcome: Bioavailability (F) of Mircera in Pediatric Participants Based on Population PK Model
Description: Bioavailability (F) is defined as the percentage of the administered drug, that reaches the systemic circulation. A population PK model was developed for Mircera that adequately describes pediatric data: a 1-compartment model with first order absorption and elimination processes. The bioavailability (F) was estimated using all the data points listed under time frame using the population PK model.
Time Frame: Pre-dose at Week 1, 9, 17; Post-dose at Week 3, Week 19 and additional sample taken between 24 hours and 5 days at participant's convenience
Population: PK population included all participants enrolled in the study.
Measure: Number; unit: percentage
Arm/Group | Mircera
Number analyzed (Participants) | 40
percentage | 67

ADVERSE EVENTS:
Time Frame: Up to Week 45
Description: Safety population included all participants who received at least one dose of study drug regardless of whether they withdrew prematurely or not.
Arm/Group | Mircera
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 13/40
Other Adverse Events (participants affected / at risk) | 28/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mircera (N=40)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Device related thrombosis (General disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (2)
Enterovirus infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 3 (3)
Pharyngotonsillitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Device malfunction (Product Issues) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mircera (N=40)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (4)
Injection site pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 5 (5)
Bronchitis (Infections and infestations) | 2 (2)
Conjunctivitis (Infections and infestations) | 3 (3)
Gastroenteritis (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (3)
Rhinitis (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 6 (6)
Urinary tract infection (Infections and infestations) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (6)
Haematuria (Renal and urinary disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hypertension (Vascular disorders) | 2 (3)
Hypotension (Vascular disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/93/NCT03552393/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT03552393/SAP_001.pdf